CLINICAL TRIAL: NCT00165399
Title: Docetaxel, Estramustine and Short Term Androgen Withdrawal for Patients With a Rising PSA After Definitive Local Treatment
Brief Title: Docetaxel, Estramustine and Short Term Androgen Withdrawal for Patients With a Rising PSA After Local Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Mary-Ellen Taplin, MD, Associate Professor of Medicine, HMS, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-230; NCT00003915 (obsolete NCT alias)
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Last update posted 2018-06-25 (Actual); Status verified 2018-06

CONDITIONS: Adenocarcinoma of the Prostate; Prostate Cancer
Keywords: Prostate cancer; PSA level; docetaxel; estramustine; hormone therapy; androgen withdrawal
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Docetaxel; Estramustine; bicalutamide; Goserelin

INTERVENTIONS:
Drug: Docetaxel — Given intravenously on day 2 of four three-week cycles
Drug: Estramustine — Taken orally three times a day for 5 days starting on day one of each three-week cycles (4 cycles)
Drug: Casodex — Started 3 weeks after last chemotherapy treatment; taken orally once a day for 15 months
Drug: Zoladex — Started one week after the start of casodex; zolades is given as an injection (in the stomach once every 3 months for a total of 5 injections.

SUMMARY:
The purpose of this study is to see if the combination of chemotherapy drugs and drugs to suppress testosterone (hormone therapy) is effective in controlling early prostate cancer.

This study will attempt to:

* stop or slow the growth of disease
* gain information about prostate cancer
* evaluate the effectiveness and side effects of the study drug

DETAILED DESCRIPTION:
* Patients will receive two medications; docetaxel and estramustine. Estramustine will be taken orally three times daily for 5 days starting on day one. Docetaxel will be given intravenously on day 2. These two drugs will be repeated every 3 weeks for a total of 4 cycles (12 weeks).
* Patients will also take dexamethasone for three days at the beginning of each cycle to help decrease the risk of side effects.
* Patients will also take coumadin every day for three months while on the chemotherapy to reduce the risk of blood clots.
* After 12 weeks the chemotherapy phase will be completed and patient will start on the hormone therapy part of the treatment. Three weeks after the last chemotherapy treatment, patients will start Casodex orally once daily.
* After taking Casodex for 1 week, patients will then start on Zoladex (an injection in the abdomen) every 3 months for a total of 5 injections.
* During study treatment various blood tests will be performed to watch the disease. Study treatment will stop after a total of 18 months (3 months chemotherapy and 15 months hormone therapy). A physical exam and blood tests will be performed every 3 months for 2 years, every 4 months for the third year, and then every 6 months after that.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented adenocarcinoma of the prostate
* Previous treatment with either radical prostatectomy or radiation therapy
* Post prostatectomy: PSA rising on at least two successive occasions at least two weeks apart
* Post radiation therapy alone: PSA has to be rising as documented on two successive occasions at least two weeks apart and also have doubled from the nadir post treatment value
* ECOG performance status 0-1
* ANC > 1,500/mm3
* Platelet counts > 100,000/mm3
* SGOT and/or SGPT may be up to 2.5 x ULN

Exclusion Criteria:

* Documented local recurrence of prostate cancer or documented metastatic disease
* History of other malignancy within the last 5 years, other than curatively treated basal cell carcinoma of the skin
* Medical condition requiring the use of concommitant corticosteroids
* Active infection
* Significant cardiac disease, angina pectoris or myocardial infarction within six months
* Prior chemotherapy including estramustine, suramin
* Active thrombophlebitis or history of thromboembolic events in the six months preceding study treatment
* Clinically significant neuropathy
* Elevated bilirubin above ULN

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-03 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2005-12-31 (Actual)

PRIMARY OUTCOMES:
To determine the feasibility of administering chemotherapy and medical castration to men with rising PSA after radical prostatectomy or radiation therapy. | 2 years

SECONDARY OUTCOMES:
To determine the PSA response rate and duration of response
to measure testosterone, free testosterone, and sex hormone binding globulin in relation to chemotherapy and hormone therapy. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mary-Ellen Taplin, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (5):
- United States (5):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic-Burlington, Burlington, Massachusetts
  - University of Massachusetts Memorial Medical Center-University Campus, Worcester, Massachusetts
  - Norris Cotton Cancer Center, Lebanon, New Hampshire